CLINICAL TRIAL: NCT04690738
Title: Role of Pancreatic Exocrine Secretion in Weight Gain After Pancreas Transplantation
Status: Suspended | Type: Observational
Why Stopped: Currently lack of funding and study staff
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20052109
Record Dates: First submitted 2020-07-31; First posted 2020-12-31 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Exocrine Pancreatic Insufficiency; Weight Gain
Keywords: pancreas transplant; weight gain; pancreatic insufficiency; kidney pancreas transplant
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post Pancreas Transplant Patients: Pancreas transplant recipients
  Interventions: Diagnostic Test: Fecal Elastase Concentration

INTERVENTIONS:
Diagnostic Test: Fecal Elastase Concentration — Stool sample for fecal elastase-1 (FEC) analysis and microbiome for sequencing and analysis will be obtained pre- and post-transplant.

SUMMARY:
Pancreas transplantation is currently the most reliable method for glycemic control in insulin dependent diabetic patients. Outcomes of pancreas transplantation have improved significantly over the years due to improved surgical techniques, medical management and immunosuppression. However, weight gain after pancreas transplantation remains a common problem with associated consequences such as development of type 2 diabetes, coronary artery disease, graft loss, metabolic syndrome and increased risk of cardiovascular death. Excessive weight gain is well known after liver and kidney transplantation; however there are very few studies that have looked at weight gain after pancreas transplantation. In a recent study by Knight et al, 26% of the pancreas transplant recipients had excessive weight gain, defined as more than 30% of their baseline weight by 1-year post transplant. The study focused mainly on the endocrine function of the pancreas, explaining that excessive peripheral insulin circulation post-transplant may explain the weight gain. Other factors like immunosuppression, increased oral intake and potentially reduced activity may also have played a role. However no study has looked at the possible role of exocrine secretion from the new pancreatic allograft, combined with exocrine secretion of the old pancreas, leading to excessive availability of digestive juices like trypsin, chymotrypsin, lipase, amylase, gelatinase, elastase etc. Our hypothesis is that the excessive weight gain after pancreas transplant, which is more than in other solid organ transplants, is driven by the excessive digestive juice leading to improved conversion of available food and nutrient into storable energy and subsequently leading to weight gain. The patient will therefore need to either increase physical activity to avoid weight gain post-transplant or significantly reduce caloric intake.

Fecal elastase test (FE-1)-elastase is a proteolytic enzyme produced by pancreatic acinar cells. They bind to bile salt and pass through the gut without degradation. These levels correlate well with the other pancreatic enzyme levels. Fecal elastase concentration (FEC) has been used routinely to screen for pancreatic exocrine insufficiency (PEI).

Exocrine pancreatic juice has been a target for the management of obesity lately, with the use of drugs like Orlistat (Xenical) that inhibits pancreatic lipase and therefore interfere with the absorption of fat. If our theory of excessive pancreatic juice availability after pancreas transplant can be proven, it can help guide the targeted use and appropriate dosing of such drugs based on the level of the pancreatic juice as measured by the FEC.

DETAILED DESCRIPTION:
This is the second of a two-part study. The first part, a pilot study, assessed the FEC level after pancreas transplant to determine if FEC is high compared to that of the general population and see if particularly high levels correlate with post pancreas transplant weight gain. The pilot study demonstrated excessively high FEC relative to the general population/healthy individuals, and much higher than the upper limit of the assay. However, the study did not show correlation between weight gain and high post-transplant FEC. This is thought to be because majority of the subjects enrolled were years from their transplant and the high FEC and weight gain already occurred early post-transplant. The study showed that FEC level was particularly high early post-transplant and decreased gradually over the years. It also showed that most weight gain occurred between years

1 to 2 post-transplant; we therefore felt the pilot study might have missed the period when the high level of exocrine secretion contributed to the weight gain. The primary aim of this second part is to assess patients from pre-transplant period to post-transplant period and see if FEC early posttransplant correlates with weight gain, particularly during the period of post-transplant weight gain established from results of the pilot study. The relationship between obesity and the gut microbiome is still not well established. To understand the role of gut microbiome in pancreas transplant patients, we will assess gut microbiome and other gut factors that may help us determine if the weight gain is related to lifestyle changes or it is associated with pancreas transplant.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of pancreas transplant with or without other organs
* Age 18 - 80 yrs

Exclusion Criteria:

* Unwillingness to consent or participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recipients of pancreas transplant with or without kidney transplant
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of Fecal Elastase-1, measured in mcg/g, correlation with post-transplant weight | Follow-up for up to 3 years post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Oyedolamu Olaitan, MBBS, Principal Investigator — Rush University Medical Center; Amanda Van Jacobs, MS, Study Director — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knight RJ, Islam AK, Pham C, Graviss EA, Nguyen DT, Moore LW, Kagan A, Sadhu AR, Podder H, Gaber AO. Weight Gain After Simultaneous Kidney and Pancreas Transplantation. Transplantation. 2020 Mar;104(3):632-639. doi: 10.1097/TP.0000000000002862. PMID 31335775
- [Background] Ewald N, Raspe A, Kaufmann C, Bretzel RG, Kloer HU, Hardt PD. Determinants of Exocrine Pancreatic Function as Measured by Fecal Elastase-1 Concentrations (FEC) in Patients with Diabetes mellitus. Eur J Med Res. 2009 Mar 17;14(3):118-22. doi: 10.1186/2047-783x-14-3-118. PMID 19380282
- [Background] Dominguez-Munoz JE, D Hardt P, Lerch MM, Lohr MJ. Potential for Screening for Pancreatic Exocrine Insufficiency Using the Fecal Elastase-1 Test. Dig Dis Sci. 2017 May;62(5):1119-1130. doi: 10.1007/s10620-017-4524-z. Epub 2017 Mar 17. PMID 28315028
- [Background] Forsmark C, Adams PC. Pancreatic function testing--valuable but underused. Can J Gastroenterol. 2009 Aug;23(8):529-30. doi: 10.1155/2009/464326. No abstract available. PMID 19668794
- [Result] Van Jacobs A, Williams MD, Ralph OG, Becerra AZ, Chan EY, Olaitan O. Pancreatic Exocrine Secretion and Weight Gain After Pancreas Transplantation. Prog Transplant. 2023 Sep;33(3):236-241. doi: 10.1177/15269248231189877. Epub 2023 Jul 30. PMID 37518975